CLINICAL TRIAL: NCT07392593
Title: Physical Activity as a Non-Invasive Strategy to Address Obesity and Musculoskeletal Risk in First-Year University Students: A Cross-Sectional Study in Spain
Status: Completed | Type: Observational
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, DeAsís-Fernández, Francisco, Director, Universidad Rey Juan Carlos
Other Study IDs: URJC-PA-OBMSK-2023
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Physical Inactivity; Sedentary Behavior; Obesity & Overweight
Keywords: Physical Activity; Sedentary Behavior; Obesity; Musculoskeletal Health
MeSH Terms: conditions — Sedentary Behavior; Obesity; Overweight; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this retrospective cross-sectional study was to assess physical activity and sedentary behavior levels in first-year university students and to explore their association with obesity and musculoskeletal health risk indicators. Physical activity and sedentary behavior were assessed using the Global Physical Activity Questionnaire (GPAQ), while body mass index (BMI) was used to classify weight status. Sedentary behavior was interpreted as an indirect indicator of musculoskeletal risk. Understanding these behavioral patterns may help identify at-risk profiles and inform non-invasive prevention strategies in university populations.

DETAILED DESCRIPTION:
Physical inactivity and prolonged sedentary behavior are recognized risk factors for obesity and musculoskeletal health problems, particularly in young adults exposed to long periods of sitting during academic activities. University students represent a population vulnerable to lifestyle-related health risks during the transition to higher education.

This retrospective observational study analyzed previously collected data from first-year university students enrolled at Universidad Rey Juan Carlos between September 2023 and June 2024. Physical activity and sedentary behavior were assessed using the Global Physical Activity Questionnaire (GPAQ), which evaluates activity across work, transportation, and leisure domains. Body mass index was calculated from self-reported height and weight and classified according to World Health Organization criteria.

The primary objective of the study was to describe physical activity and sedentary behavior patterns and to examine their associations with obesity and indirect indicators of musculoskeletal risk. No intervention, treatment, randomization, or follow-up procedures were performed as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* First-year university students enrolled at Universidad Rey Juan Carlos
* Availability of complete GPAQ data

Exclusion Criteria:

* Incomplete GPAQ data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First-year university students enrolled at Universidad Rey Juan Carlos, Madrid (Spain)
Sampling Method: Non-Probability Sample
Enrollment: 821 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level (Total MET-minutes per week) | Retrospective assessment during the academic year 2023-2024
  Physical activity assessed using the Global Physical Activity Questionnaire (GPAQ), including work, transportation, and leisure domains. Total physical activity was expressed as MET-minutes per week.

SECONDARY OUTCOMES:
Sedentary Behavior | Retrospective assessment during the academic year 2023-2024
  Self-reported daily sitting time assessed using the Global Physical Activity Questionnaire (GPAQ) and interpreted as an indirect indicator of musculoskeletal health risk.
Body Mass Index (BMI) | Retrospective assessment during the academic year 2023-2024
  Body mass index calculated as weight (kg) divided by height squared (m²) and classified according to World Health Organization criteria.
Physical Activity Risk Categories | Retrospective assessment during the academic year 2023-2024
  Classification into low, moderate, or high physical activity levels based on World Health Organization GPAQ thresholds.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Madrid, Spain